CLINICAL TRIAL: NCT07251517
Title: Cognitive Impairment Post Stroke: a Single-blinded Randomized Trial on the Efficacy of TEleRehabilitation. The CIPS-TER Study
Brief Title: Cognitive Rehabilitation in Post-stroke Cognitive Impairment
Acronym: CIPS-TER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Collaborators: University of Milan (Other); University of Pavia (Other)
Responsible Party: Principal Investigator, Anna Poggesi, Associate professor, PhD, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25546
Record Dates: First submitted 2025-10-02; First posted 2025-11-26 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Cognitive Impairment; Stroke Acute
Keywords: cognitive telerehabilitation; stroke; cognitive impairment; neuropsychology
MeSH Terms: conditions — Cognitive Dysfunction; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive telerehabilitation treatment (Experimental): The cognitive telerehabilitation program will be based on the Virtual Reality Rehabilitation System (VRRS) of the Khymeia group (Noventa Padovana, Italy). The VRRS equipment includes a central workstation located in the clinical center and VRRS tablet devices used independently by patients to perform cognitive exercises. The cognitive modules of the VRRS include a broad set of tasks for each major cognitive domain. Tasks can be customized and supervised from the central workstation and comprehensive automatic reports are available for each rehabilitation session.
  Interventions: Procedure: Cognitive telerehabilitation treatment
- Standard Care (No Intervention): Participants in the control group, "standard care", will be instructed to have a usual lifestyle and will receive conventional treatments and clinical indications provided by referring doctors.

INTERVENTIONS:
Procedure: Cognitive telerehabilitation treatment — The subjects who will be part of the experimental group will receive a total of up to 40 hours of individual treatment. Cognitive telerehabilitation will be administered in five weekly sessions of 60 minutes each for a total of 8 weeks. The cognitive treatment will include twenty-four exercises aimed at improving memory, attention, executive functions and visuospatial skills. In each treatment session, participants will work with six exercises, lasting 10 minutes each, and the difficulty of the task will increase adaptively over the course of the home sessions.
  Arms: Cognitive telerehabilitation treatment

SUMMARY:
The goal of this 2-year, prospective, single-blind randomized clinical trial is to investigate: the efficacy in reducing the risk of cognitive impairment 6 months after stroke; the generalizability of cognitive reinforcement to real life, such as activities of daily living and quality of life; and the impact on cognitive performance. In the treatment group, feasibility, adherence, and satisfaction with the cognitive telerehabilitation program will also be evaluated. Participants will be adult patients with a diagnosis of ischemic or hemorrhagic stroke, within 5-21 days after onset.

The main outcomes to be evaluated are:

* diagnosis of cognitive impairment (primary outcome);
* activities of daily living, quality of life, changes in frailty status, and cognitive efficiency (secondary outcomes).

There will be two groups: a treatment group and a control group. Participants in the treatment group will undergo a cognitive telerehabilitation program of 40 hours over 8 weeks, while participants in the control group will be instructed to follow their standard care.

DETAILED DESCRIPTION:
Despite its social and economic burden, cognitive impairment after stroke is still a neglected consequence compared to other neurological deficits for which rehabilitation pathways are routinely available. Cognitive telerehabilitation represents an emerging, promising and innovative approach that has the potential to provide both an individualized treatment and the opportunity of access to services for a wide catchment area.

CIPS-TER study is a 2-year prospective, single-blind, randomized clinical trial. A cognitive telerehabilitation program, versus standard care, will be administered to a cohort of stroke patients with the aims to investigate: efficacy in reducing the risk of cognitive impairment 6 months after stroke; generalizability of the cognitive reinforcement to real life, such as activities in daily living and quality of life; and impact on cognitive performances. In the treated group, feasibility, adherence and appreciation of the cognitive telerehabilitation program will also be evaluated. During an enrolment period of 12 months, all adult patients consecutively admitted to Stroke Unit of Careggi University Hospital and/or to Intensive Rehabilitation Unit of IRCCS Don Gnocchi in Florence with a diagnosis of ischemic or hemorrhagic stroke will be evaluated, within 5-21 days after onset, for the inclusion in the study.

After baseline assessment, the foreseen cohort of 100 enrolled patients will be randomly assigned to treatment or control group. The cognitive telerehabilitation program (Virtual Reality Rehabilitation System, Khymeia) will consist of up to 40 hours (8 weeks) of individual treatment based on memory, attention and executive functions, and visuospatial tasks to be to autonomously performed with a tablet. All patients will be followed after 2 months (brief cognitive assessment) and after 6 months (comprehensive clinical, functional, and cognitive assessment). The study outcomes will be evaluated at 6-month follow-up visit and will include the diagnosis of cognitive impairment (primary outcome), and activities of daily living, quality of life, changes in frailty status and cognitive efficiency (secondary outcomes). The results of CIPS-TER study will contribute to our knowledge on the potentials of an early cognitive telerehabilitation on the reduction of persistent cognitive and functional burden in stroke patients, and thus on the utility to consider cognitive telerehabilitation as an effective component of post-stroke care pathways. In line with precision medicine, CIPS-TER project could also help to highlight which clinical features characterize those stroke patients that could maximally benefit of such cognitive interventions. Finally, experiences and setups gathered within CIPS-TER project could represent a technical and methodological background for future studies aimed at the development and/or the evaluation of cognitive telerehabilitation systems in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of ischemic or hemorrhagic stroke between 5 and 21 days after the event
* Ability to express written informed consent
* Evidence of impairment of global cognitive efficiency according to the post-stroke MoCA (MoCA total score≤21)
* Normal stenia of at least one upper limb (NIHSS motor item of at least one upper limb=0)

Exclusion Criteria:

* Pre-existing dementia (IQ-CODE>3.48 and/or diagnosis of dementia by a specialist).
* Severe aphasia (NIHSS language item ≥2 and impaired performance on the Token test, i.e. a correct score below the 5th centile of the normal population).
* Withdrawal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Reduction of the risk of cognitive impairment post stroke in the medium-long term | From enrollment to 6 months after stroke
  The primary endpoint will be the diagnosis of cognitive impairment, which will include both mild cognitive impairment (MCI) and dementia and will be made according to the DSM-5 criteria for the diagnosis of mild or major neurocognitive disorders, respectively.

SECONDARY OUTCOMES:
Quality of life post-stroke | From enrollment to 6 months after stroke
  Secondary endpoint will be quality of life post-stroke. Quality of life measured by means of the Stroke-adapted sickness impact profile (SA-SIP) scale and EuroQol visual scale (score 0-100). In the SA-SIP scale high scores indicate a strong impact of the disease. To calculate the score, the items must be weighted, added up for each subscale, and expressed as a percentage for each subscale from 0 to 100%. As regards EuroQOL, high scores mean better outcomes.
Independence in activities of daily living post-stroke | From enrollment to 6 months after stroke
  Another secondary endpoint will be independence in activities of daily living post-stroke. Functional status measured by means of the Activities of Daily Living scale (ADL) Instrumental Activities of Daily Living scale (IADL). ADL score 0-6, IADL score 0-22. Higher scores mean a better outcome.
Changes in frailty status post-stroke | From enrollment to 6 months after stroke
  Another endpoint will be changes in frailty status post-stroke. Frailty measured according to the Italian version of the Tilburg Frailty Indicator (TFI). The TFI is an easy and simple to administer self-report questionnaire developed to evaluate frailty in community-dwelling older adults (Total score 0-15:). Each patient that will obtain a total score 5 will be classified as frail. Higher scores mean worse outcome.
Impact on cognitive performance | From enrollment to 6 months after stroke
  Another endpoint will be impact on cognitive performance and changes in cognitive efficiency. Cognitive performances at the multidomain neuropsychological battery will be compared between telerehabilitation and standard care groups in order to evaluate a potential treatment benefit on the overall cognitive profile. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florence, Florence, Firenze, Italy